CLINICAL TRIAL: NCT00731328
Title: HLA-HAPLOIDENTICAL FAMILIAL DONOR HEMATOPOIETIC CELL TRANSPLANTATION AFTER REDUCED INTENSITY CONDITIONING OF BUSULFAN, FLUDARABINE, AND ANTI-THYMOCYTE GLOBULIN FOR PATIENTS WITH BONE MARROW FAILURE SYNDROME - A PHASE 2 STUDY
Brief Title: Donor Stem Cell Transplant After Busulfan, Fludarabine, Methylprednisolone, and Antithymocyte Globulin in Treating Patients With Bone Marrow Failure Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Kyoo-Hyung Lee, Professor of Internal Medicine, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000600351; AMC-UUCM-2008-0038
Record Dates: First submitted 2008-08-08; First posted 2008-08-11 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Nonmalignant Neoplasm; Paroxysmal Nocturnal Hemoglobinuria
Keywords: refractory anemia; refractory anemia with ringed sideroblasts; refractory cytopenia with multilineage dysplasia; childhood myelodysplastic syndromes; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; aplastic anemia; paroxysmal nocturnal hemoglobinuria
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Neoplasms; Hemoglobinuria, Paroxysmal; Anemia, Refractory; Anemia, Aplastic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation — infusion of mobilized donor hematopoietic progenitor cells

SUMMARY:
RATIONALE: Giving low doses of chemotherapy and antithymocyte globulin before a donor stem cell transplant helps stop the growth of abnormal cells. It may also stop the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining abnormal cells (graft-versus-tumor effect).

PURPOSE: This phase II trial is studying how well a donor stem cell transplant works after busulfan, fludarabine, methylprednisolone, and antithymocyte globulin in treating patients with bone marrow failure syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the efficacy of HLA-haploidentical familial donor hematopoietic stem cell transplantation after reduced-intensity conditioning regimen comprising busulfan, fludarabine phosphate, and anti-thymocyte globulin in patients with bone marrow failure syndromes.

OUTLINE:

* Reduced-intensity conditioning regimen: Patients receive busulfan IV daily on days -7 and -6, fludarabine phosphate IV over 30 minutes on days -7 to -2, anti-thymocyte globulin (ATG) IV over 4 hours on days -4 to -1, and methylprednisolone IV over 30 minutes starting 30 minutes before ATG on days -4 to -1.
* HLA-haploidentical donor hematopoietic stem cell transplantation: Patients receive donor hematopoietic stem cells via Hickman catheter over 1 hour on days 0 or 1.
* Graft-versus-host-disease prophylaxis (GVHD): Patients receive cyclosporine IV over 2-4 hours every 12 hours starting on day -1 (cyclosporine can be given orally once oral medication can be tolerated) and methotrexate IV on days 2, 4 , 7, and 12. In the absence of GVHD, cyclosporine is tapered starting between days 30 to 60.

After completion of study treatment, patients are followed periodically for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of any of the following bone marrow failure syndromes:

  * Severe aplastic anemia, meeting 1 of the following criteria:

    * Not responsive to immunosuppressive therapy
    * With recurrent cytopenia after immunosuppressive therapy or allogeneic hematopoietic cell transplantation
  * Low-risk myelodysplastic syndrome, including any of the following:

    * Refractory anemia
    * Refractory anemia with ringed sideroblasts
    * Refractory cytopenia with multi-lineage dysplasia
  * Paroxysmal nocturnal hemoglobinuria, meeting 1 of the following criteria:

    * With thrombotic episodes
    * With severe cytopenia
* No willing, suitable HLA-compatible donor in family or in donor registries

  * Related donor with HLA-haploidentical mismatch at three or less of 6 loci
  * Patients with very severe neutropenia (< 200/μL) or febrile episodes, who feel urgent need for allogeneic hematopoietic cell transplantation, are eligible without a search for HLA-matched unrelated donors

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Bilirubin < 2.0 mg/dL
* AST < 3 times upper limit of normal
* Creatinine < 2.0 mg/dL
* Ejection fraction > 40% by MUGA scan

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Donor cell engraftment | 10-35 days after transplantation
  neutrophil count over 500/ul

SECONDARY OUTCOMES:
Regimen-related toxicities as assessed by NCI's Common Toxicity Criteria | 0-60 months after transplantation
  various toxicities of treatment
Acute and chronic GVHD | 15-100 days; 100 days to 4 years
  ocurrence of acute or chronic GVHD after transplantation
overall survival | 0-60 months
  patients surviving after transplantaion
event-free survival | 0-60 months after transplatation
  patients undergoing transplantation and maintaining donor hematopoiesis

CONTACTS AND LOCATIONS:
Overall Officials: Kyoo H. Lee, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center - University of Ulsan College of Medicine, Seoul, South Korea